CLINICAL TRIAL: NCT05775250
Title: Evaluation of Giomer Varnish Versus Fluoride Varnish on The Color Improvement of White Spot Lesions in Permanent Teeth of Children: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Two Varnishes on the Improvement of White Spot Lesions in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Naglaa Ibrahim Ezz, Associate professor, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-D 262-3
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: White Spot Lesion
Keywords: white spot lesion; fluoride varnish; Giomer Varnish

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- giomer varnish (Experimental): Giomer varnish containing surface pre-reacted glass-ionomer (PRG) filler, will be administrated once.
  Interventions: Drug: giomer varnish
- fluoride varnish (Active Comparator): 5% NaF fluoride varnish, it will be administrated once.
  Interventions: Drug: giomer varnish

INTERVENTIONS:
Drug: giomer varnish — Giomer varnish containing surface pre-reacted glass-ionomer (PRG) filler, will be administrated once.

SUMMARY:
A randomized control trial evaluating the effect of the Giomer varnish versus fluoride varnish on the color improvement of the white spot lesion in permanent anterior teeth of children aged between 8-14 years by using a spectrophotometer at baseline, after 1 month, 3 months and 6 months

ELIGIBILITY:
Inclusion Criteria:

* • Patients with good general health.

  * Adequate oral hygiene,
  * Patients who didn't receive remineralizing agents during the last 3 months other than regular toothpaste.

Exclusion Criteria:

* Uncooperative child.
* Active carious lesion.
* Labial surface restoration.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
white spot lesion color change | 6 months
  assessment of white spot lesion color by using spectrophotometer

SECONDARY OUTCOMES:
Patient response to the treatment | 6 months
  Patient response to the treatment using facial image scale, scores from 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa I Ezzeldin, Ass. Prof, Principal Investigator — October University for Modern Sciences and arts, Cairo, Egypt
Locations (1):
- October University of Modern Sciences and Arts, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided